CLINICAL TRIAL: NCT02145013
Title: Assessment and Impact of Portal Hypertension Before and During Liver Resection in Patients With Hepatocellular Carcinoma
Brief Title: Portal Hypertension and Liver Resection in Patients With Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Chetana LIM, MD, Henri Mondor University Hospital
Other Study IDs: LIM Chetana
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Primary Liver Cancers
Keywords: portal hypertension, hepatocellular carcinoma, resection
MeSH Terms: conditions — Hypertension, Portal; Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Portal hypertension: Hepatectomy
  Interventions: Procedure: Liver resection
- No portal hypertension: Hepatectomy
  Interventions: Procedure: Liver resection

INTERVENTIONS:
Procedure: Liver resection — Hepatectomy by either open, laparoscopic or robotic procedures

SUMMARY:
According to the BCLC guidelines, surgical resection of hepatocellular carcinoma complicating cirrhosis is restricted to patients with preserved liver function, single nodule without vascular invasion and with hepatic venous gradient below 10 mmHg.

However, other guideline treatment, especially from eastern countries demonstrated that surgical resection is safe and feasible and provides better survival than the treatment recommended by the BCLC system for patients with similar stage.

The primary goal of this study is to assess the impact of HVPG on short and long-term outcomes in HCC patients who undergo liver resection.

DETAILED DESCRIPTION:
Patients with HCC and candidates for hepatectomy are classified into two groups according to the presence of portal hypertension. Short- and long-term outcomes will be compared.

ELIGIBILITY:
Patients with hepatocellular carcinoma who undergo surgical resection (intention to treat analysis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with hepatocellular carcinoma
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-12 (Actual); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 90 day
  In-hospital or 90-day mortality

SECONDARY OUTCOMES:
morbidity | 90 day
  Overall and liver-related complications including liver failure, ascites, biliary fistula, bleeding, pulmonary complications, and renal complications.
  Grading system according to Clavien-Dindo classification
Survival outcomes | 1,3 and 5 years
  Including Overall survival and disease free survival

OTHER OUTCOMES:
Acute kidney injury | within 90 days after surgery
  As defined by the KDIGIO criteria
Sarcopenia | Before liver resection
  using computed tomography
Time from diagnosis to liver resection | from the date of diagnosis until the date of first referral and from the date of first referral to date of hepatectomy, assessed up to 3 months
Impact of PET CT on overall survival following liver resection | Before liver resection
  quantitative assessment of metabolic uptake (FDG and choline)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Azoulay, MD PhD, Principal Investigator — Henri Mondor
Locations (1):
- Henri Mondor University Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ishizawa T, Hasegawa K, Aoki T, Takahashi M, Inoue Y, Sano K, Imamura H, Sugawara Y, Kokudo N, Makuuchi M. Neither multiple tumors nor portal hypertension are surgical contraindications for hepatocellular carcinoma. Gastroenterology. 2008 Jun;134(7):1908-16. doi: 10.1053/j.gastro.2008.02.091. Epub 2008 Mar 8. PMID 18549877
- [Derived] Lim C, Salloum C, Chalaye J, Lahat E, Costentin CE, Osseis M, Itti E, Feray C, Azoulay D. 18F-FDG PET/CT predicts microvascular invasion and early recurrence after liver resection for hepatocellular carcinoma: A prospective observational study. HPB (Oxford). 2019 Jun;21(6):739-747. doi: 10.1016/j.hpb.2018.10.007. Epub 2018 Nov 3. PMID 30401520
- [Derived] Lim C, Osseis M, Lahat E, Doussot A, Sotirov D, Hemery F, Lanteri-Minet M, Feray C, Salloum C, Azoulay D. Safety of laparoscopic hepatectomy in patients with hepatocellular carcinoma and portal hypertension: interim analysis of an open prospective study. Surg Endosc. 2019 Mar;33(3):811-820. doi: 10.1007/s00464-018-6347-1. Epub 2018 Jul 12. PMID 30003350
- [Derived] Lim C, Salloum C, Osseis M, Lahat E, Gomez-Gavara C, Compagnon P, Luciani A, Feray C, Azoulay D. Short-term outcomes following hepatectomy for hepatocellular carcinoma within and beyond the BCLC guidelines: A prospective study. HPB (Oxford). 2018 Mar;20(3):222-230. doi: 10.1016/j.hpb.2017.08.027. Epub 2017 Sep 19. PMID 28935451